CLINICAL TRIAL: NCT02211079
Title: An Open-Label, Fixed-Sequence Study in Healthy Male Subjects to Assess the Drug Interaction Potential of Multiple-Doses of JNJ-54861911 With a Drug "Cocktail" Representative for CYP3A4, CYP2B6, CYP2C9, and CYP1A2 Substrates
Brief Title: A Study to Assess Effect of JNJ-54861911 on Pharmacokinetics of Cocktail Representatives for Cytochrome P450 (CYP) 3A4, CYP2B6, CYP2C9, and CYP1A2 Substrates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR105152; 54861911ALZ1010 (Other: Janssen Research & Development, LLC); 2014-001794-14 (EudraCT Number)
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Healthy; JNJ-54861911; Caffeine; Midazolam; Tolbutamide; Cytochrome P450 3A4; Cytochrome P450 2C9; Cytochrome P450 1A2; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — atabecestat; Caffeine; Midazolam; Tolbutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JNJ-54861911 + Caffeine + Midazolam +Tolbutamide (Experimental): JNJ-54861911, 50 milligram (mg) (2*25 mg tablets) orally once daily from Day 2 to Day 9 along with caffeine 100 mg (2*50 mg tablets), midazolam 2 mg (1 milliliter [mL], 2 mg/mL solution), and tolbutamide 500 mg tablet, orally on Day 1, 2, and 9.
  Interventions: Drug: JNJ-54861911; Drug: Caffeine; Drug: Midazolam; Drug: Tolbutamide

INTERVENTIONS:
Drug: JNJ-54861911 — JNJ-54861911, 50 mg (2*25 mg tablets) orally once daily from Day 2 to Day 9.
Drug: Caffeine — Single oral dose of caffeine 100 mg (2*50 mg tablets), on Day 1, 2, and 9.
Drug: Midazolam — Single oral dose of midazolam 2 mg (1 mL, 2 mg/mL solution), on Day 1, 2, and 9.
Drug: Tolbutamide — Single oral dose of Tolbutamide 500 mg tablet, on Day 1, 2, and 9.

SUMMARY:
The purpose of this study is to assess the effects of single and multiple once daily doses of 50 milligram (mg) of JNJ-54861911 on pharmacokinetics (PK) (study of the way a drug enters and leaves the blood and tissues over time) of caffeine, midazolam, and tolbutamide in healthy male participants.

DETAILED DESCRIPTION:
This is a single-center, open-label (participants and researchers are aware about the treatment, participants are receiving), fixed-sequence study in healthy male participants. The study consists of 3 phases: Screening Phase (within 21 to 2 days prior to the first dose administration on Day 1), Open Label Treatment Phase (Day 1 up to Day 9), and Follow-up Phase (7 to 14 days after discharge from the study unit on Day 10 or at early withdrawal). The maximum duration of study will be 7 weeks per participant. During the Open-Label Treatment Phase, participants will receive JNJ-54861911, 50 mg (2*25 mg tablets) orally once daily from Day 2 to Day 9 along with caffeine 100 mg (2*50 mg tablets), midazolam 2 mg (1 milliliter [mL], 2 mg/mL solution), and tolbutamide 500 mg tablet, orally on Day 1, 2, and 9. Blood samples will be collected pre-dose (Day 1) up to Day 10 to understand the PK characteristics of midazolam, 1-hydroxy midazolam (midazolam metabolite), caffeine, paraxanthine (caffeine metabolite), tolbutamide, 4-hydroxytolbutamide and carboxytolbutamide (tolbutamide metabolites). In addition, a blood sample will be collected on Day -1 from all enrolled participants to study genetic factors that may influence the PK, safety, and/or tolerability of JNJ-54861911 and co-medications. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study, and are willing to participate in the study
* Body mass index between 18 and 30 kilogram per square meter
* Must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening or admission (up to Day 1 pre-dose)
* Man, who is sexually active with a woman of child-bearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the Investigator, and must also agree to not donate sperm during the study and for 90 days after receiving the last dose of study drug
* Participant must be healthy on the basis of clinical laboratory tests performed at Screening as per Investigator's judgment

Exclusion Criteria:

* History of or current liver or renal insufficiency, closed-angle glaucoma, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, dermatological or metabolic disturbances
* Known allergies, hypersensitivity, or intolerance to JNJ-54861911 or its excipients, sulfonamides, midazolam, caffeine or tolbutamide.
* History of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening
* History of drug or alcohol abuse according to current Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria within 6 months before Screening or positive test result(s) for alcohol and/or drugs of abuse (including barbiturates, opiates, cocaine, cannabinoids, amphetamines, metamphetamines, benzodiazepines and cotinine) at Screening or admission
* Smoking of cigarettes (or equivalent) and/or used nicotine based products within 3 months prior to study drug administration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Pre-dose on Day 1,2,3,9,10 and 0.5,1,1.5,2,2.5,3,4,6,8,10,12,16 hours post-dose on Day 1,2,9 (for Caffeine and Tolbutamide); Pre-dose on Day 1,9 and 0.5,1,1.5,2,2.5,3,4,6 hours post-dose on Day 1,2,9 (for Midazolam)
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Concentration (Tmax) | Pre-dose on Day 1,2,3,9,10 and 0.5,1,1.5,2,2.5,3,4,6,8,10,12,16 hours post-dose on Day 1,2,9 (for Caffeine and Tolbutamide); Pre-dose on Day 1,9 and 0.5,1,1.5,2,2.5,3,4,6 hours post-dose on Day 1,2,9 (for Midazolam)
  The Tmax is time to reach the maximum observed plasma concentration.
Time to Last Quantifiable Plasma Concentration (Tlast) | Pre-dose on Day 1,2,3,9,10 and 0.5,1,1.5,2,2.5,3,4,6,8,10,12,16 hours post-dose on Day 1,2,9 (for Caffeine and Tolbutamide); Pre-dose on Day 1,9 and 0.5,1,1.5,2,2.5,3,4,6 hours post-dose on Day 1,2,9 (for Midazolam)
  The Tlast is time to last observed quantifiable plasma concentration (Clast).
Area Under the Plasma Concentration-time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Pre-dose on Day 1,2,3,9,10 and 0.5,1,1.5,2,2.5,3,4,6,8,10,12,16 hours post-dose on Day 1,2,9 (for Caffeine and Tolbutamide); Pre-dose on Day 1,9 and 0.5,1,1.5,2,2.5,3,4,6 hours post-dose on Day 1,2,9 (for Midazolam)
  The AUC (0-last) is area under the plasma concentration-time curve from time zero to time of last quantifiable concentration.
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0 - infinity]) | Pre-dose on Day 1,2,3,9,10 and 0.5,1,1.5,2,2.5,3,4,6,8,10,12,16 hours post-dose on Day 1,2,9 (for Caffeine and Tolbutamide); Pre-dose on Day 1,9 and 0.5,1,1.5,2,2.5,3,4,6 hours post-dose on Day 1,2,9 (for Midazolam)
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to extrapolated infinite time, calculated as the sum of AUC (0-last) and Clast/lambda(z), where AUC (0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time; Clast is the last observed quantifiable concentration; and lambda(z) is first-order rate constant associated with the terminal portion of the semilogarithmic drug concentration-time curve.
Area Under the Plasma Concentration-time Curve From Time Zero to Time 24 Hours (AUC [0-24]) | Pre-dose on Day 1,2,3,9,10 and 0.5,1,1.5,2,2.5,3,4,6,8,10,12,16 hours post-dose on Day 1,2,9 (for Caffeine and Tolbutamide); Pre-dose on Day 1,9 and 0.5,1,1.5,2,2.5,3,4,6 hours post-dose on Day 1,2,9 (for Midazolam)
  The AUC (0-24) is area under the plasma concentration-time curve from time zero to time 24 hours.
Elimination Half-Life (t1/2) | Pre-dose on Day 1,2,3,9,10 and 0.5,1,1.5,2,2.5,3,4,6,8,10,12,16 hours post-dose on Day 1,2,9 (for Caffeine and Tolbutamide); Pre-dose on Day 1,9 and 0.5,1,1.5,2,2.5,3,4,6 hours post-dose on Day 1,2,9 (for Midazolam)
  Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve, is calculated as 0.693 divided by lambda(z), where lambda(z) is first-order rate constant associated with the terminal portion of the curve. The t1/2 is the measure of time, for plasma concentration to decrease by one half.
Elimination Rate Constant (lambda[z]) | Pre-dose on Day 1,2,3,9,10 and 0.5,1,1.5,2,2.5,3,4,6,8,10,12,16 hours post-dose on Day 1,2,9 (for Caffeine and Tolbutamide); Pre-dose on Day 1,9 and 0.5,1,1.5,2,2.5,3,4,6 hours post-dose on Day 1,2,9 (for Midazolam)
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the semilogarithmic drug concentration-time curve.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Baseline up to follow-up (7 to 14 days after discharge from the study unit on Day 10 or at early withdrawal)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Groningen, Netherlands